CLINICAL TRIAL: NCT00850304
Title: Feasibility Study of Treatment of Non Promyelocytic Acute Myeloid Leukaemia on Elderly Patients by Low Dose Cytosar Plus Arsenic Trioxide on Ambulatory Schedule
Brief Title: Treatment of Non Promyelocytic Acute Myeloid Leukaemia on Elderly Patients by Low Dose Cytosar Plus Arsenic Trioxide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Mahdi Jalili M.D., Hematology-Oncology and SCT Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87-02-36-7242
Record Dates: First submitted 2009-02-21; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm one (Experimental)
  Interventions: Drug: Cytosar; Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Cytosar — Cytosar 20 mg /q12h/ sc/10d/q28d for 2 cycle
Drug: Arsenic trioxide — Arsenic trioxide 10mg/infusion2h/iv/DW5% d1-d5,d7-d11
  Other Names: ATO

SUMMARY:
Our purpose in this study is to explore the feasibility of treatment of non promyelocytic Acute myeloid leukaemia on elderly patients. We select ten patients with age further than 60 with comorbidity and treat by low dose cytosar subcutaneous plus arsenic trioxide for ten days in month. We will assess overall response rate and overall survival in end of one year.

DETAILED DESCRIPTION:
Acute myeloid leukemia is a disease in which characterised by blast further than 20% in bone marrow plus incomplete differentiation. Many of this patients are elderly with age further than 60 years(CALGB,ECOG,EORTC) or 55 years (SWOG). Mortality rate fallowing standard therapy of this patients is high that can reach to 50%. One of methods to apply a remission with least mortality and morbidity and also significant lower cost effects compare to historical and conventional standard regimen is low dose cytosar and arsenic trioxide combination that has been reported complete remission to 34%.

We select ten patients with age further than 60 with comorbidity and treat by low dose cytosar subcutaneous plus arsenic trioxide for ten days in month. We will assess overall response rate and overall survival in end of one year.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients with non promyelocytic AML
* Performance status (ECOG) 3 or 4

Exclusion Criteria:

* Age <60 years
* Elevation of AST OR ALT more than ten times above normal
* Serum bilirubin above 5
* Cr level > 2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Response Rate | 1, 2, 6 month and one year after intervention

SECONDARY OUTCOMES:
Overall Survival | One year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Alimoghaddam, M.D., Study Director — Hematology-Oncology and SCT Research Center
Locations (1):
- Hematology-Oncology and SCT Research Center, Tehran, Tehran Province, Iran